CLINICAL TRIAL: NCT04904484
Title: A Safety Assessment of the iZephyr Hood for Non Invasive Ventilation in COVID-19 Patients
Brief Title: A Safety Assessment of the iZephyr Hood for NIV in COVID-19 Patients
Acronym: iZephyr
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Mercedes AMG PETRONAS Formula One Team (Unknown); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 292573
Record Dates: First submitted 2021-04-15; First posted 2021-05-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Aerosol Disease; Covid19; Noninvasive Ventilation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Environmental contamination of SARS Co-V2 (air and surface) will be tested around COVID patients receiving Non-invasive ventilation or high flow oxygen therapy before using the iZephyr hood and then with the iZephyr hood in place, to determine if the hood changes the amount of environmental contamination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With i-zephyr (Experimental): using the hood
  Interventions: Device: iZephyr hood
- Without i-zephyr (No Intervention): Not using the hood

INTERVENTIONS:
Device: iZephyr hood — Assessment of an aerosol containment device
  Arms: With i-zephyr

SUMMARY:
This study is a safety assessment of the iZephyr hood a novel aerosol removal device in patients receiving non invasive ventilation for COVID-19.

DETAILED DESCRIPTION:
Demonstrate that safety and suitability of the iZephyr Hood in patients receiving non-invasive ventilation (NIV) or high flow oxygen therapy (HFOT).

Determine the user acceptability of the iZephyr Hood in patients receiving NIV and HFOT.

Determine the reduction in aerosol spread of COVID-19 viral particles when using the Zephyr hood in patients using non-invasive ventilation or high flow oxygen.

ELIGIBILITY:
Inclusion Criteria:

Adult COVID-19 negative patients who are requiring non-invasive ventilation (phase II)

Adult COVID-19 positive patients who are requiring non-invasive ventilation (Phase III)

Exclusion Criteria:

Patients under the age of 18 years or those lacking capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Determine the background concentration of SARS-Co-V2 around COVID patients receiving NIV | 3 month
  Air and surface sampling for SARS Co-V2 around COVID patients receiving non invasive ventilation or high flow oxygen therapy.
Determine the background concentration of SARS-Co-V2 when the iZephyr hood is in use | 12 months
  Air and surface sampling for SARS Co-V2 around COVID patients receiving non invasive ventilation or high flow oxygen therapy inside an iZephyr hood.
Impact of iZephyr hood on environmental SARS Co-V2 contamination | 12 months
  Determine if there is a change in the concentration of SARS-Co-V2 virus on the surfaces and in the air samples surrounding a COVID-19 positive patient whilst using the iZephyr compared to when not using the iZephyr.

IPD SHARING:
Plan to Share IPD: No